CLINICAL TRIAL: NCT01285219
Title: A Multicenter, Randomized, Cross-over Phase 3 Comparing Preventive Pegylated Filgrastim and Filgrastim in Cancer Patients Receiving Myelosuppressive Chemotherapy
Brief Title: A Study Comparing Pegylated Filgrastim and Filgrastim in Support for Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Beijing Chest Hospital (Other); Hospital affiliated to Academy of Military Medical Sciences (Unknown); Tianjin Medical University Cancer (Unknown); Fudan University (Other); First Hospital of China Medical University (Other); Hunan Cancer Hospital (Other); West China Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Peking University Third Hospital (Other); Tianjin People's Hospital (Other); Qilu Hospital of Shandong University (Other); Zhejiang Cancer Hospital (Other); Changhai Hospital (Other)
Responsible Party: Dr. Yuankai Shi, Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, 100021, China
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PEG3; 2002SL0047 (Registry Identifier: State Food and Drug Administration of China)
Record Dates: First submitted 2011-01-24; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Cancer
Keywords: Granulocyte colony-stimulating factor , recombinant; Polyethylene glycols; Neutropenia; Drug therapy, combination
MeSH Terms: conditions — Neoplasms; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AOB,pegylated filgrastim to filgrastim (Active Comparator): patients were administered pegylated filgrastim 100 ug/kg in cycle 1 and ﬁlgrastim 5 ug/kg/d in cycle 2
  Interventions: Drug: pegylated filgrastim and ﬁlgrastim
- BOA,ﬁlgrastim to pegylated filgrastim (Active Comparator): patients received ﬁlgrastim 5 ug/kg/d in cycle 1 and pegylated filgrastim 100 ug/kg in cycle 2
  Interventions: Drug: ﬁlgrastim and pegylated filgrastim

INTERVENTIONS:
Drug: pegylated filgrastim and ﬁlgrastim — patients were administered pegylated filgrastim 100 ug/kg in cycle 1 and ﬁlgrastim 5 ug/kg/d in cycle 2
  Arms: AOB,pegylated filgrastim to filgrastim
Drug: ﬁlgrastim and pegylated filgrastim — patients received ﬁlgrastim 5 ug/kg/d in cycle 1 and pegylated filgrastim 100 ug/kg in cycle 2
  Arms: BOA,ﬁlgrastim to pegylated filgrastim

SUMMARY:
Neutropenia is one of the most frequent adverse effects of chemotherapy, and the main factor to limit the dosage and delay the schedule of chemotherapy. Preventive filgrastim administration has long been established as the standard of care. A pegylated filgrastim was independently developed by GeneLeuk Biopharmaceutical Co., Ltd, Shandong, China. It composed of filgrastim and a 20 kd polyethylene glycol molecule covalently bound at the N-terminal residue. Preclinical studies phase 1 and phase 2 trials have shown that pegylated filgrastim has decreased renal clearance, increased plasma half-life, and prolonged efficacy in compare with ﬁlgrastim. These characters were similar to those of Neulasta.

The investigators designed a multicenter, randomized, cross-over phase Ⅲ trial to compare the efficacy and safety of a single injection of pegylated filgrastim and daily injections of ﬁlgrastim in chemotherapy naive patients receiving commonly used regimens. The hypothesis is that pegylated filgrastim is similarly effective and safe with regular filgrastim.

DETAILED DESCRIPTION:
This was a multicenter, randomized, open-label, cross-over, noninferiority study to evaluate whether a single injection of pegﬁlgrastim is as effective and safe as daily injections of ﬁlgrastim in patients receiving commonly used chemotherapy regimens. Patients were randomly assigned in a 1:1 ratio to AOB and BOA arm with center as the stratiﬁcation variables. All the patients received two cycles of chemotherapy of identical regimen and dosage. In arm AOB, patients were administered pegylated filgrastim 100 ug/kg in cycle 1 and ﬁlgrastim 5 ug/kg/d in cycle 2; while in arm BOA, patients received ﬁlgrastim 5 ug/kg/d in cycle 1 and pegylated filgrastim 100 ug/kg in cycle 2.

Study drugs Both filgrastim and pegylated filgrastim were provided by GeneLeuk Biopharmaceutical Co., Ltd, Shandong, China.

In cycle 1 of AOB arm and cycle 2 of BOA arm, on 9 am of day 3, patients were to receive a dose of 100µg/kg of pegylated filgrastim, based on actual body weight, as a single s.c. injection.

In cycle 2 of AOB arm and cycle 1 of BOA arm, patients were to receive daily s.c. injection of filgrastim at a dose of 5 µg/kg/day. Injections began on 9 am of day 3 and continued daily until an absolute neutrophil count (ANC) ≥10.0 × 109 /l was documented after the expected nadir or for a maximum of 14 days, whichever occurred first.

Chemotherapy Treatment All cytotoxic agents were administrated on day 1 of the 21-day regimens. The regimens include PC(paclitaxel 175 mg/m2; carboplatin area under curve[AUC] 5～6 or cisplatin 75 mg/m2 )； AC (doxorubicin [or pirarubicin]60 mg/m2 or epirubicin 100 mg/m2；cyclophosphamide 600 mg/m2), PA(paclitaxel 175 mg/m2 ；doxorubicin [or pirarubicin]50 mg/m2 or epirubicin 80 mg/m2）； CHOP (cyclophosphamide 750mg/m2；doxorubicin[or pirarubicin] 50 mg/m2 or epirubicin100 mg/m2；vincristine1.4 mg/m2；prednisone 100mg，po，day 1-5)。 Efficacy measurements Blood samples were collected for complete blood counts (cbc) with differential on days 0, 3, 5, 7, 9, 11, 13, 17 and 21 of each cycle. Day 0 was defined as the day before day one, in cycle 1 it is the base line, and in cycle 2 is day 21 of cycle 1.

The primary efficacy end point was protective rate of grade 4 neutropenia after chemotherapy (defined as the rate of ANC keeps above 0.5 × 109 /l through the whole cycle). The secondary efficacy end points included the rate of grade 3/4 neutropenia, time to neutrophil recovery (deﬁned as the time from chemotherapy administration until the patient's ANC increased to 2.0 × 109/l after the expected nadir), incidence of febrile neutropenia (defined as ANC<0.5×109/L and auxiliary temperature>38.0℃), incidence of antibiotic administration and ANC profile.

Safety assessments Patients recorded their auxiliary temperature daily, and were monitored for adverse events throughout the study. Before chemotherapy and in the third week of each chemotherapy cycle, serum hepatic and renal function, electrolysis, urine routine test and electrocardiograph were examined.

The safety endpoint of this study was incidence and severity of adverse events (WHO grade 1-4), side effects, and changes in clinical laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of malignant solid tumours (excluding highly aggressive lymphomas such as lymphoblastic lymphoma and Burkitt lymphoma)
* chemotherapy naive
* Karnofsky Performance Status ≥70
* age 18-70 years; normal white blood cell (WBC) count and platelet count
* adequate renal, hepatic and cardiac function
* life expectancy ≥3 months
* normal bone marrow function

Exclusion Criteria:

* history of systematic chemotherapy (including adjuvant therapy)
* large area radiotherapy (>25% of bone marrow volume)
* uncontrolled infection
* bone marrow involvement
* pregnancy, lactation
* history of blood stem cell or organ transplantation
* antibiotic administration within 72 hours of enrolment
* long time exposure to glucocorticoids and immunosuppressive agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2006-01; Primary Completion 2007-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Protective rate of grade 4 neutropenia | 21 days
  the rate of ANC keeps above 0.5 × 109 /l through the whole cycle

SECONDARY OUTCOMES:
rate of grade 3/4 neutropenia | 21 days
  the rate of ANC lower than 1.0 × 109 /l
time to neutrophil recovery | 21 days
  the time from chemotherapy administration until the patient's ANC increased to 2.0 × 109/l after the expected nadir
incidence of antibiotic administration | 21 days
  rate of using antibiotic in a cycle
ANC profile | 21 days
  the dynamic change of ANC number
incidence and severity adverse events | 21 days
  unexpected and untoward events
incidence and severity of side effects | 21 days
  expected and untoward events caused by study drug or control drug
changes in clinical laboratory values | 21 days
  changes in clinical laboratory values
incidence of febrile neutropenia | 21 days
  rate of ANC<0.5×109/L and auxiliary temperature>38.0℃

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D., Principal Investigator — Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, 100021, China

REFERENCES:
- [Derived] Yang S, He X, Liu P, Zhou S, Dong M, Qin Y, Yang J, Zhang C, Han X, Shi Y. [Duration of filgrastim prophylaxis for chemotherapy-induced neutropenia and its predictors]. Zhonghua Zhong Liu Za Zhi. 2016 Jan;38(1):69-72. doi: 10.3760/cma.j.issn.0253-3766.2016.01.013. Chinese. PMID 26796810